CLINICAL TRIAL: NCT01985620
Title: The Impact of a Short Intervention During RSV Prophylaxis on Influenza Vaccination Rate and Morbidity in Infants Born Premature.
Brief Title: The Impact of a Short Intervention During RSV Prophylaxis on Influenza Vaccination Rate.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-13-YS-0503-13-CTIL; 0503-13-TLV
Record Dates: First submitted 2013-11-10; First posted 2013-11-15 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2013-11

CONDITIONS: Prematurity; RSV; Influenza; Upper Respiratory Tract Infection; Lower Respiratory Tract Infection
Keywords: Vaccination; RSV; Influenza; Prematurity
MeSH Terms: conditions — Premature Birth; Influenza, Human; Respiratory Tract Infections | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Active Comparator): Educational intervention with the parents
  Interventions: Behavioral: Educational intervention
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational intervention
  Arms: study group

SUMMARY:
Premature infants (born before 34 wk) are routinely vaccinated against RSV but vaccination rate against influenza are low in spite of national programs. Study goal is to evaluate the effectiveness of short intervention during RSV prophylaxis visit, planned to educate parents about the importance of influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Infants coming for RSV prophylaxis

Exclusion Criteria:

* Already vaccinated against influenza
* Contraindication for influenza vaccination

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination rate | 5 months

SECONDARY OUTCOMES:
respiratory morbidity | 5 months
  Upper and lower respiratory tract events during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel